CLINICAL TRIAL: NCT01441089
Title: Collection of Blood From Therapeutic Trial Participants for Analysis of Genetic Differences in Drug Disposition and Pharmacokinetics of Probe Medications
Brief Title: Collection of Blood From Patients With Cancer, Other Tumors, or Tumor Predisposition Syndromes for Genetic Analysis
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110242; 11-C-0242
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Prostate Cancer; Breast Cancer; Lung Cancer; Ovarian Cancer; Lymphoma
Keywords: Pharmacogenetics; Pharmacokinetics; Pharmacodynamics; Clinical Outcome; Drug Metabolism and Transport; Natural History; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Ovarian Neoplasms; Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Patients with cancer, other tumors, or possible genetic tumor: Patients enrolled on IRB approved NIH Intramural Research Program (IRP) therapeutic clinical trials

SUMMARY:
Background:

- Some genes may be associated with a greater chance of side effects during cancer treatment. These genes may also make certain treatments less effective. Researchers want to collect blood or cheek swab samples from people having cancer treatment to study these genes.

Objectives:

- To obtain a blood or cheek swab sample to study genetic differences that may affect cancer treatment.

Eligibility:

- Individuals with cancer who are being treated at the National Cancer Institute.

Design:

* Participants will provide a blood sample for study.
* Participants who have blood-based cancer, such as leukemia, will provide a cheek swab sample.
* If the blood or cheek swab sample does not have enough genetic material for analysis, an additional sample may be collected.

DETAILED DESCRIPTION:
Background:

* Genetic polymorphisms in drug-metabolizing enzymes, transporters/receptors might affect an individual's response to drug therapy.
* Inter-individual differences in efficacy and toxicity of antitumor agents are especially important given the narrow therapeutic index of these drugs.
* During analysis of investigational agents, inter-individual variation in pharmacokinetics (PK) and pharmacodynamics (PD) is most often noted. Genetic variation in genes encoding proteins that regulate or mediate the metabolism and transport of drugs often account for some of the wide variation seen in PK/PD, and ultimately the response to, and toxicity from, pharmaceutical agents.
* The administration of probe substrates can be used to determine the phenotype of enzymes and transporters responsible for drug disposition, providing a useful tool to better understand the cause of unexpected AEs or toxicities of clinical trial participants.

Objectives:

-Explore potential associations between genetic variants discovered with Pharmacoscan involved in inter-individual differences in drug disposition versus the pharmacokinetics, pharmacodynamics of pharmaceutical agents.

Eligibility:

-Any individual currently enrolled on IRB approved NIH Intramural Research Program (IRP) therapeutic clinical trials.

Design:

* Exploratory study with a planned accrual of 1,100 participants.
* Genomic DNA extracted from blood samples collected from participants (participants with leukemia will have cheek swab samples collected) will be analyzed.
* In cases where participants carry genetic variants that related to poor outcome or significant toxicity on a given drug, clinical recommendations will be provided where specific instructions are available in the package insert.
* The association between variants in Pharmacoscan-covered genes will be correlated with PK/PD and clinical outcomes such as response and/or toxicity.
* Genotyping and/or phenotyping probe administration will be used to identify potential genetic variants with unknown or poorly defined drug interactions, including genetic variants with unknown metabolic phenotype and drugs with poorly defined metabolic pathways in the literature.
* The Clinical Pharmacology Program (CPP) will measure the plasma concentration of enzyme or transporter phenotyping probe substrates (or send the sample out to a third party if the assay is commercially available) in select participants enrolled on clinical trials at the CCR.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any individual currently enrolled in an NIH intramural research program clinical trials receiving treatment.
* Ability of participant or Legally Authorized Representative (LAR) to understand and be willing to sign the informed consent document.
* Age >= 3 years old

EXCLUSION CRITERIA:

-N/A

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient enrolled on an IRB approved NIH Intramural Research Program therapeutic clinical trial with cancer, other tumors, or possible genetic tumor predisposition syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2012-05-21 (Actual)

PRIMARY OUTCOMES:
Obtain and analyze the genomic DNA from patients with cancer, other tumors, or possible genetic tumor predisposition syndromes on a therapeutic clinical trial. | duration of study
  to determine the association between SNP parameters and clinical response and/or toxicity from genomic DNA extracted from patient samples

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-C-0242.html